CLINICAL TRIAL: NCT07362277
Title: The Effect of Mat Pilates on Body Composition and Physical Activity Levels in Sedentary Women Emerging Adulthood
Brief Title: Mat Pilates on Body Awareness and Physical Activity Levels in Sedentary Emerging Adulthood Women
Acronym: mat pilates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, MUSA ÇANKAYA, Dr. MUSA ÇANKAYA, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUSA CANKAYA,
Record Dates: First submitted 2025-12-23; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Exercise Therapy; Awareness; Sedentary Behavior; Woman's Role; Exercise
Keywords: Exercise Therapy; Awareness; Sedentary Behavior; Woman's Role; Exercise
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: Posttest and Control Group Randomize Controlled
Who Masked: Participant
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-Pilates training (experimental) group (Experimental): Participants in our study will be divided into two groups. Group 1: The Pilates training (experimental) group will undergo 8 weeks of Pilates exercise training, 3 times a week, for an average of 1 hour. Pilates exercises include pelvic exercises, chest movements (breathing exercises), leg movements to strengthen the lower extremities, flight movements, core exercises, pendulum exercises, and cat-cow exercises, which will be performed by participants in the exercise group. The exercises will be:
  • Roll-up, Roll-over, Single-leg circle, Rolling like a ball, Single-leg stretch, Double-leg stretch, Spinal stretch, Swinging with legs apart. After 2 weeks, they will be made a little more challenging.
  Interventions: Other: Pilates training (experimental)
- 2-Control Group (No Intervention): The other 27 participants will be assigned to the control group. An initial assessment will be conducted, followed by a second assessment after 8 weeks.

INTERVENTIONS:
Other: Pilates training (experimental) — Pilates training
  Other Names: Pilates training
  Arms: 1-Pilates training (experimental) group

SUMMARY:
This study investigating the effects of mat pilates on body awareness and physical activity levels in sedentary women transitioning to adulthood, 27 control groups and 27 mat pilates exercise groups will be included. The groups will be compared at the end of an 8-week exercise program. Participants' socio-demographic characteristics, body awareness (using the Body Awareness Questionnaire), and physical activity level (using the Tegner Physical Activity Questionnaire and the International Physical Activity Questionnaire short-form scales) will be assessed.

DETAILED DESCRIPTION:
The World Health Organization (WHO) recommends physical activities of varying intensity tailored to different age groups. Evidence shows that regular physical activity reduces the risk of various chronic diseases such as heart attack, cerebrovascular accident, diabetes, and cancer, and positively impacts overall health by improving mental health and quality of life. Pilates is one of the popular and widespread physical activities that can be recommended worldwide. There are different classifications of this exercise form, such as classical, modern, and clinical (modified) Pilates. Pilates is a physical method and holistic approach that provides mental focus and reduces stress and anxiety. Pilates exercise was founded by Joseph Pilates in the 1920s. The traditional principles of Pilates exercise include centering, concentration, control, precision, flow, and breathing. The Pilates method focuses on exercises that involve breath control, postural symmetry, and the stabilization and flexibility of the spine, pelvis, and shoulders. Participation in Pilates exercises has been shown to correct poor posture, strengthen muscles that affect poor posture, maintain body balance, and thus alleviate spinal deformities. Emerging adulthood (for women) refers to the life stage between the end of adolescence and the onset of stable adulthood. In high-income countries, this refers to the ages of 18-29. While development during this period shares many similarities with the preceding period of adolescence and the subsequent period of young adulthood, emerging adulthood exhibits some significant differences in terms of demographics, subjective aspects, and identity exploration. This is a period of independence and exploration, but it can also be accompanied by stress and anxiety. Therefore, while there are important opportunities to lay a solid foundation for a healthy adulthood, mental health problems and psychiatric disorders are common at this life stage. People face significant life and role changes during this period, such as entering and leaving educational settings, leaving home, starting a career, and finding a life partner [5]. Emerging adulthood (i.e., late adolescence and early adulthood, ages 18-30) is characterized by five distinct features: Identity exploration: the emerging adult asks, "Who am I?" They try to find an answer to the question and evaluate various options, instability that can arise in interpersonal relationships or different environments (work, home, etc.), self-focus where the emerging adult makes their own decisions and learns to be self-sufficient, a transitional period between adolescence and adulthood and a feeling between possibilities/optimism, the hope that everything is possible and everything can be achieved. At this developmental stage, for individuals, discovering themselves and others and the new feelings that this can awaken can sometimes make it difficult to maintain harmonious relationships and sometimes conflicts can arise, which can turn into attacks of intimate partner violence.

A sedentary lifestyle is associated with the development of chronic noncommunicable diseases, increased mortality rates, and mental health disorders characterized by symptoms of depression and anxiety. Regular physical activity offers various benefits in terms of cardiovascular, respiratory, metabolic, musculoskeletal, functional health, cancer prevention, various chronic noncommunicable diseases, and mental health. However, research shows that children and adolescents who engage in higher levels of physical activity experience better physical health, mental, and psychosocial well-being compared to those with a sedentary lifestyle.

In health studies, developing body awareness has been shown to be a therapeutic approach for chronic pain, obesity, and post-traumatic stress disorder. Body awareness involves attention and awareness of internal bodily sensations, contributes to physical balance and well-being, and is linked to body image. Emotional regulation and sense of self are associated with physical sensations linked to emotions. It is influenced by awareness. Body awareness is linked to the subjective and phenomenological aspects of proprioception and interoception, which contribute to consciousness and are shaped by mental processes such as attention, interpretation, evaluation, beliefs, memories, conditioning, attitudes, and emotions. Therefore, body awareness emerges from the interaction of neurological and behavioral aspects, the environment, and the individual's psychomotor structure.

A review of the literature reveals that there are few studies on women in the transition to adulthood. Furthermore, there is insufficient information on how sedentary women's body awareness and physical activity levels change with Pilates. Our study was designed to examine the effects of mat Pilates on body awareness and physical activity levels in sedentary women in the transition to adulthood.

ELIGIBILITY:
Inclusion Criteria:

* Possess the ability to read and understand Turkish, be between the ages of 18 and 29,
* I have a sedentary lifestyle, possess the cognitive ability to understand and interpret survey questions, and for sedentary participants, not have engaged in regular exercise for 2 months, have a Physical Activity Score (IPAQ) -short form of less than 600 Metabolic Equivalent of Task (MET) minutes per week, and body weight below 130 kg.

Exclusion Criteria:

* Participants with chronic, neurological, orthopedic, rheumatic systemic and/or lung disease, those who exercise/sport, have a history of malignancy, are pregnant, have a history of fracture in the last year,
* I have chronic kidney or liver disease, have cardiovascular disease, and have peripheral vestibular disorder were excluded.

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 54 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Body Awareness Survey | 1 assessment before exercise, 1 assessment after exercise (8 weeks).
  Developed in 1989, the BAS is a measure that assesses an individual's sensitivity to normal or abnormal physical states and processes, incorporating physical, emotional, and social elements, and questioning sensitivity to physical reactions . The BAS [8] has been found to be the measure with the best performance. Participants were asked to rate each of the 18 statements on a scale of 1 to 7 (1 = Not true for me at all, 7 = Very true for me). The total score from the questionnaire can be 126 or at least 18. Rating in the questionnaire is based on the total score. The higher the score, the better the level of body awareness.
Tegner Activity Survey (TAS) | 1 assessment before exercise, 1 assessment after exercise(8 weeks).
  TAS is scored on a scale of 0-10 based on daily living and sports activities. There are 11 activity levels on this scale. It determines patients' activity levels by inquiring about their daily living activities, leisure activities, or competitive sports. On this scale, level 0 represents complete disability, level 4 represents participation in recreational activities, and level 10 represents elite athletes.
International Physical Activity Questionnaire - Short Form (IPAQ-SF) | 1 assessment before exercise, 1 assessment after exercise (8 weeks).
  UFAA-KF aims to compare the physical activity levels of individuals aged 18-65 over the past week. The long form of the questionnaire consists of 27 items that allow for a detailed assessment of housework, occupational activity, gardening, transportation, and leisure activities. The short form of the questionnaire consists of 7 items that determine the time spent walking, sitting, and engaging in moderate and vigorous activities. The UFAA-KF, consisting of seven questions that collect information about the time participants spent on vigorous physical activity, moderate physical activity, walking, and sitting in the past week, was tested for validity and reliability in Turkish. Participants' metabolic equivalent of task (MET) values are calculated as follows .

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Seydişehir Health Services Vocational School, Therapy and Rehabilitation Department, Konya, Tyrkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided